CLINICAL TRIAL: NCT03912597
Title: Reducing Stigma Against Depression: Designing and Implementing a VR-assisted Curriculum to Reduce Students' Perceptions of Patients With Depression
Brief Title: VR-assisted Curriculum on Depression for Stigma Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-18-208
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Control; Behavior
Keywords: virtual reality; stigma reduction; depression; mental health campaigns; user experience; enjoyment; presence
MeSH Terms: conditions — Behavior; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality [A] (Experimental): Participants watch a 4-minute virtual reality video, on top of reading a brochure, then answer post-intervention questionnaires.
  Interventions: Device: Virtual Reality; Device: Brochure
- Brochure Waitlist Control [A] (Active Comparator): Participants read an informational brochure about depression, then answer post-intervention questionnaires. After that, they will be given a chance to watch the VR video at the end of their participation session.
  Interventions: Device: Brochure
- Standard Video Control [B] (Active Comparator): Participants watch a 4-minute standard video. After which, using a video, a discussion of the video will be facilitated for participants to contextualise and understand the video better. Then, participants answer post-intervention questionnaires.
  Interventions: Device: Brochure; Device: Standard Video Control
- Virtual Reality [B] (Experimental): Participants answer pre-questionnaires, then watch a 4-minute virtual reality video. After which, using a video, a discussion of the video will be facilitated for participants to contextualise and understand the video better. Then, participants answer post-intervention questionnaires.
  Interventions: Device: Virtual Reality; Device: Brochure

INTERVENTIONS:
Device: Virtual Reality — The 4-minute virtual reality video depicts a day in a life of a student with depression. The one-take video, filmed with a 360° camera, is designed to provide users with an immersive experience that simulates what it feels like to have depression. The user interface consisted of a Google Cardboard VR headset attached to a smartphone.
  Arms: Virtual Reality [A]; Virtual Reality [B]
Device: Brochure — Participants read an informational brochure about depression depicting standard information about depression, including symptoms and information on how to support someone with depression.
Device: Standard Video Control — The 4-minute standard video depicts a similar storyline as was shown in the VR video. The standard video is filmed from a third-party perspective with multiple takes edited into a final video, following the standard filming style of these videos. The standard video will be viewed from a laptop with headphones attached.
  Arms: Standard Video Control [B]

SUMMARY:
Two randomised controlled trials will be conducted to evaluate a virtual reality (VR) simulation designed to reduce stigma against depression. Qualitative interviews will also be carried out to evaluate the VR simulation.

DETAILED DESCRIPTION:
The investigators examine the impact of a VR-assisted curriculum on stigma reduction towards individuals with depression. This is done through the development and evaluation of a VR-assisted curriculum that promotes stigma reduction towards depression among tertiary-aged students. Collection of data will provide insights about the effectiveness of VR's immersive quality in enhancing stigma reduction skills through measures of attitudes, beliefs and knowledge about depression. In the first study, VR is compared with traditional pamphlets in an information sharing booth about depression. In the second study, participants attend a 30-min session where they undergo an educational curriculum with either a VR or standard video as adjunctive tools.

ELIGIBILITY:
Inclusion Criteria:

* Tertiary students from NUS and Yale-NUS only

Exclusion Criteria:

* History of medical or psychiatric disorder; History of motion sickness, dizziness or epilepsy; (For reliability and safety of heart-rate monitoring) Tattoos near the wrist and/or nickel or acrylate allergies

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
Stigmatising beliefs towards depression | 2 minutes
  The extent of agreement with negative beliefs and stereotypes about depression will be adapted from the 10-item agreement sub-scale of the Self-Stigma of Mental Illness Scale.
Stigmatising attitudes towards depression | 5 minutes
  Stigmatising attitudes refer to the opinions that one has towards persons with depression, and how they would interact with these group of people. This will be measured using an adapted version of the Attribution Questionnaire-27.
Knowledge about depression | 2 minutes
  A Depression Literacy measure will be used to assess participants' understanding and knowledge of depression.
Video Enjoyment | 1 minute
  In the VR condition, enjoyment of the VR simulation will be assessed through five items on a video enjoyment questionnaire created by the researchers, that includes items such as "I found the video interesting" and "The video made me more interested in the topic" on a visual analog scale. The scale was anchored between 0 indicating "Strongly Disagree" to 10 indicating "Strongly Agree".
Video Presence | 1 minute
  Presence felt in the VR simulation will be assessed through four items on a video presence questionnaire, that includes items such as "How aware were you of events happening in your actual surroundings outside of the video?" and "How strong was your sense of 'being there' in the video environment?" on a visual analog scale. The questions were adapted from the original Presence Questionnaire by Witmer and Singer (1998) that outlined four sub-factors of control, sensory, distraction and realism; items in our questionnaire were carefully selected to represent all of the factors. The scale ranged from 0 indicating "Not At All" to 10 indicating "Very Much So".

SECONDARY OUTCOMES:
Affect (PANAS) | 3 minutes
  Participants' mood will be assessed using the Positive and Negative Affect Scale (PANAS) as a secondary measure of user experience with the respective videos. The PANAS consists of two 10-item subscales assessing positive and negative affect, and is rated on a 5-point scale ranging from 1 representing "Very Slightly or Not at All" to 5 representing "Extremely".
Heart rate live tracking | 4 minutes
  Changes in heart rate, assessed live during the video viewing duration, will be measured as a physiological measure of user experience.
Qualitative feedback about VR video | 10 minutes
  Participants will be invited to give feedback on their VR experience. Questions in the qualitative interview will address (1) their thoughts on mental health awareness amongst the public, (2) their experience watching the VR simulation and (3) reasons for stopping, or not, at similar mental health booths with VR simulations in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore